CLINICAL TRIAL: NCT00189839
Title: A Multicentre, Randomised, Double Blind, Two Arm Parallel Group Study to Evaluate and Compare the Efficacy and Safety of Modified Release Tacrolimus FK506E (MR4) Versus Tacrolimus FK506 in Combination With MMF (Cellcept®) and Steroids in Patients Undergoing Kidney Transplantation
Brief Title: A Study to Evaluate the Safety and Efficacy of FK506E (MR4) in Patients Undergoing Primary Kidney Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Disclosure Office Europe, Astellas Pharma Europe BV
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FG-506E-12-03
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Kidney Transplantation
Keywords: Tacrolimus; Kidney transplantation; Transplantation, kidney; Renal Transplantation; Transplantation, renal
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: tacrolimus
- 2 (Experimental)
  Interventions: Drug: tacrolimus

INTERVENTIONS:
Drug: tacrolimus — Immunosuppression
  Other Names: FK506E, MR4

SUMMARY:
The purpose of this study is to evaluate and to compare the efficacy and safety of a triple modified release tacrolimus FK506E (MR4) / MMF / steroid regimen with a triple standard tacrolimus FK506 / MMF / steroid regimen in patients undergoing kidney transplantation. It shall be demonstrated that FK506E (MR4) is non-inferior to FK506 with regards to the primary endpoint.

DETAILED DESCRIPTION:
A multicentre, 1:1 randomised, double blind, double dummy, two arm parallel group phase III study comparing a triple modified release tacrolimus FK506E (MR4) / MMF / steroid regimen with a triple standard tacrolimus FK506 / MMF / steroid regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving a kidney transplant from a cadaveric donor or a living non HLA identical donor between 5 and 65 years of age with compatible ABO blood type.
* Patients with end stage kidney disease who are suitable candidates for primary renal transplantation or re-transplantation (unless the graft was lost because of immunological reasons within 12 months).

Exclusion Criteria:

* Patients receiving or having previously received an organ transplant other than a kidney.
* Patients with a high immunological risk, defined as a panel reactive antibodies (PRA) grade >50% in the previous 6 months and/or with a previous graft survival of less than 12 months due to immunological reasons.
* Cold ischaemia time of the donor kidney >30 hours.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 699 (Actual)
Dates: Start 2004-08; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Time to and incidence of biopsy-proven acute rejections | 12 months

SECONDARY OUTCOMES:
Overall rate of acute rejections | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: B Krämer, Principal Investigator — Klinikum der Universität Regensburg
Locations (76):
- Argentina (2):
  - Buenos Aires
  - Santa Fe
- Australia (4):
  - Melbourne
  - Sydney
  - Westmead
  - Woudville South
- Innsbruck, Austria
- Belgium (2):
  - Brussels
  - Leuven
- Brazil (4):
  - Campinas - SP
  - Porto Alegre
  - Rio de Janeiro - RJ
  - San Paulo - SP
- Canada (4):
  - Halifax, Nova Scotia
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Prague, Czechia
- Helsinki, Finland
- France (10):
  - Créteil
  - Grenoble
  - Le Kremlin-Bicêtre
  - Lille
  - Montpellier
  - Nantes
  - Nice
  - Saint-Etienne
  - Toulouse
  - Vandœuvre-lès-Nancy
- Germany (10):
  - Berlin
  - Bochum
  - Cologne
  - Erlangen
  - Essen
  - Frankfurt
  - Halle
  - Hann
  - München
  - Regensburg
- Greece (2):
  - Athens
  - Thessaloniki
- Budapest, Hungary
- Dublin, Ireland
- Italy (7):
  - Bari
  - Milan
  - Padua
  - Palermo
  - Pisa
  - Siena
  - Treviso
- Mexico (2):
  - Cuernavaca Morelos
  - Mexico City
- Netherlands (2):
  - Maastricht
  - Utrecht
- Oslo, Norway
- Poland (2):
  - Bydgoszcz
  - Szczecin
- South Africa (3):
  - Cape Town
  - Durban
  - Pretoria
- Spain (8):
  - A Coruña
  - Badalona Barcelona
  - Barcelona
  - Córdoba
  - Madrid
  - Málaga
  - Santander
  - Seville
- Sweden (2):
  - Gothenburg
  - Uppsala
- Zurich, Switzerland
- United Kingdom (5):
  - Belfast
  - Birmingham
  - Coventry
  - Glasgow
  - Manchester

REFERENCES:
- [Derived] Kramer BK, Albano L, Banas B, Charpentier B, Backman L, Tedesco-Silva H Jr, Lehner F, Mondragon-Ramirez GA, Glyda M, Cassuto-Viguier E, Viklicky O, Mourad G, Rigotti P, Schleibner S, Kamar N. Efficacy of Prolonged- and Immediate-release Tacrolimus in Kidney Transplantation: A Pooled Analysis of Two Large, Randomized, Controlled Trials. Transplant Proc. 2017 Nov;49(9):2040-2049. doi: 10.1016/j.transproceed.2017.07.011. PMID 29149958